CLINICAL TRIAL: NCT01924676
Title: An Open-label, Single-dose, Randomized, Three-way Crossover Study to Estimate the Effects of Food on Oxycodone Pharmacokinetics Following Oral 40 Mg Doses of PF-00345439 Formulation K and to Estimate Its Relative Bioavailability of Oxycodone Compared to PF-003454390 Formulation X in the Fasted State in Healthy Volunteers
Brief Title: Food Effect And Relative Bioavailability Study Of Oxycodone in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pain Therapeutics (Industry)
Responsible Party: Sponsor
Organization: PainT (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B4501022
Record Dates: First submitted 2013-08-14; First posted 2013-08-16 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: food effect; pharmacokinetics; bioavailability; oxycodone; management of moderate to severe pain
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone
- Treatment B (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone
- Treatment C (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation X, single dose, under fasting conditions
  Arms: Treatment A
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation K, single dose, under fasting conditions
  Arms: Treatment B
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation K, single dose, under fed conditions
  Arms: Treatment C

SUMMARY:
To estimate the effects of food on oxycodone pharmacokinetics after administration of 40 mg doses of PF-00345439 Formulation K and to estimate its relative bioavailability compared to PF-00345439 Formulation X in the fasted state in healthy volunteers

DETAILED DESCRIPTION:
This study will estimate the effect of food (standard high-fat breakfast) on the pharmacokineticsand relative bioavailability of oxycodone following oral administration of single 40 mg doses of PF-00345439 Formulation K in healthy volunteers.

Additionally, the study will estimate the pharmacokinetics and relative bioavailability of oxycodone following oral administration of single 40 mg doses of the test PF-00345439 Formulation K compared with the reference PF-00345439 Formulation X under fasted conditions in healthy volunteers and assess the single-dose safety and tolerability of oxycodone in PF-00345439 formulations in healthy volunteers when administered under a naltrexone block.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between 18 and 55 years of age (inclusive).

Exclusion Criteria:

* Evidence or history of clinically significant disease
* Positive urine drug test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48 hours post-dose
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Maximum Observed Plasma Concentration (Cmax) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48 hours post-dose

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48 hours post-dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Concentration at time 24 hours (C24) of oxycodone, as data permit. | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48 hours post-dose
  Concentration at time 24 hours (C24) of oxycodone, as data permit.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48 hours post-dose
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Plasma Decay Half-Life (t1/2) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48 hours post-dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Baltimore, Maryland, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4501022&StudyName=Food%20Effect%20And%20Relative%20Bioavailability%20Study%20Of%20Oxycodone%20in%20Healthy%20Volunteers